CLINICAL TRIAL: NCT00165282
Title: Mindfulness Meditation in Bone Marrow Transplantation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Dana-Farber Cancer Institute (Other); University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Susan Bauer-Wu, PhD, RN, FAAN, Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IRB00005285
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Hematologic Malignancy; Bone Marrow Transplantation; Stem Cell Transplantation
Keywords: Meditation; Mindfulness meditation; Bone Marrow Transplant; Stem Cell Transplant
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Usual Care (No Intervention): Normal standard of care
- Nurse education (Active Comparator): Meets with oncology nurse
  Interventions: Behavioral: Nurse education
- Mindfulness training (Experimental): Taught Mindfulness meditation
  Interventions: Behavioral: Mindfulness training

INTERVENTIONS:
Behavioral: Mindfulness training — Taught mindfulness meditation by mindfulness instructor (trained health care professional/RN) and audio c/d
  Arms: Mindfulness training
Behavioral: Nurse education — Meets with oncology nurse to have questions answered about medical treatments and side effects
  Arms: Nurse education

SUMMARY:
The main purpose of this study is to examine techniques to help patients cope better with the stem cell/bone marrow transplant procedure.

DETAILED DESCRIPTION:
Patients will be assigned to one of three study groups:

1. receives the normal standard care;
2. meets with an oncology nurse educator, in addition to the regular nurses on the transplant team. The nurse educator will provide information and answers to patient's questions about the stem cell/bone marrow transplant experience; or
3. is taught mindfulness meditation by a nurse who is trained to be a mindfulness instructor and by an audio CD.

Mindfulness meditation is a technique that may help in coping with the stress and difficulties associated with cancer and undergoing a stem cell/bone marrow transplant. It involves learning to be in the present moment by paying attention to your breathing, sights, and sounds, and to sensations you may be experiencing, or thoughts and feelings you may be having.

Mindfulness meditation has been shown to be helpful to patients in the clinic who have cancer and other medical conditions.

Patients, regardless of random group assignment, will complete a questionnaire 8 different times, from before they are admitted to the hospital until 6 months after discharge.

Patients will also provide two urine samples while in the hospital to measure the levels of stress hormones present in the urine.

ELIGIBILITY:
Inclusion Criteria:

* Autologous stem cell transplantation for hematologic malignancy
* First transplant
* 21 years of age or older
* Speaks and understands English

Exclusion Criteria:

* Planned tandem (more than one) transplant
* Taking corticosteroids on a regular basis for a chronic condition
* Prior formal mindfulness meditation training
* Significant cognitive impairment and/or confirmed psychosis or thought disorder

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2005-04; Primary Completion 2010-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Psychological functioning | 1 year

SECONDARY OUTCOMES:
Number of days to bone marrow engraftment | 1 year
Medication use | 1 year
Urinary stress hormones (cortisol and catecholamines) | 1 year
Transplant related complications | 1 year
Hospital length of stay and re-hospitalizations | 1 year
Physical symptoms | 1 year
Quality of life | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Susan Bauer-Wu, PhD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts